CLINICAL TRIAL: NCT07199114
Title: Strength Training and Modified CrossFit in Older Adults: a Comparative Perspective
Brief Title: Crossfit in Special Population
Acronym: CrossfitUJA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CrossfitUJA
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Postural Balance; Strength Training Adaptations; Aging
Keywords: Aging;; postural balance; Strength Training Adaptations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted CrossFit Program (Experimental): Supervised, scaled functional multi-joint training tailored to older adults, combining strength and metabolic conditioning with progressive overload over 12 weeks.
  Interventions: Behavioral: Adapted CrossFit Program (12 weeks)
- Usual Activity (Control) (No Intervention): Participants maintain habitual daily activities with no structured training.

INTERVENTIONS:
Behavioral: Adapted CrossFit Program (12 weeks) — Supervised sessions focused on functional, multi-joint movements adapted for older adults; emphasis on safety and progressive overload.
  Arms: Adapted CrossFit Program

SUMMARY:
This randomized, parallel-group clinical trial evaluates a 12-week adapted CrossFit program versus usual activity in community-dwelling older adults. The primary endpoint is change in Timed Up and Go (TUG) from baseline to 12 weeks. Secondary outcomes include Functional Reach (FRT), Romberg (eyes closed), gait velocity, stride length, and lower-limb power tests (Chair-Stand, Stair Ascent, Stair Descent; time and W/kg). Sixty participants were randomized (1:1). Analyses used repeated-measures ANOVA with Bonferroni adjustments and Cohen's d effect sizes.

DETAILED DESCRIPTION:
Participants were screened and randomized (1:1) to an adapted CrossFit program (12 weeks) or to maintain usual activities (no structured training). Baseline characterization included demographics, anthropometrics, Mini-Mental State Examination (MMSE ≥ 26), physical activity level, and handgrip strength. Balance outcomes: Romberg (s, eyes closed), gait velocity (m/s), stride length (cm), TUG (s), and FRT (cm). Lower-limb power: Chair-Stand (s; W/kg), Stair Ascent/Descent (s; W/kg). Statistical analysis: normality (Shapiro-Wilk), homogeneity (Levene), repeated-measures ANOVA with Bonferroni post-hoc, and Cohen's d effect sizes. A priori sample size (G*Power 3.1): effect size 0.25, α = 0.05, power 0.80 → target n = 60 to account for attrition.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling older adults able to walk independently without assistance.

Cognitive function preserved, defined as a score of 26 points or higher on the Mini-Mental State Examination.

Absence of severe health conditions that would interfere with participation in exercise training.

Exclusion Criteria:

Presence of active neuromuscular or musculoskeletal disorders that prevent safe exercise participation.

Severe cardiovascular, pulmonary, or metabolic disease that contraindicates moderate-intensity exercise.

Any other medical or psychological condition that, in the opinion of the investigators, would make participation unsafe or unreliable.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG), seconds | Baseline and Week 12
  Change in functional mobility. Shorter time indicates better performance and reduced risk of falls.

SECONDARY OUTCOMES:
Functional Reach Test (FRT) | Baseline and 12 weeks
  Change in dynamic balance assessed by the distance a participant can reach forward without losing stability. Greater distance indicates better balance.
Chair-Stand Test (CST) | Baseline and 12 weeks
  Sit-to-stand repetitions (5 times). Lower time and higher relative power indicate better lower-limb strength and functional capacity.
Fear of Falling (Falls Efficacy Scale-International, FES-I) | Baseline and week 12
  Self-reported concern about falling during daily activities. Higher scores indicate greater fear of falling.
Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | Baseline and week 12
  Subjective sleep quality over the previous month. Higher scores indicate poorer sleep quality.
Anxiety and Depression (Hospital Anxiety and Depression Scale, HADS) | Baseline and week 12
  Symptoms of anxiety and depression measured with HADS. Higher subscale scores indicate greater severity.
Gait Velocity, meters per second | Baseline and week 12
  Walking speed measured over a standardized distance. Higher speed indicates better mobility.
Stride Length, centimeters | Baseline and week 12
  Average step length during gait assessment. Longer stride indicates better gait performance.
Kinesiophobia (Tampa Scale of Kinesiophobia, TSK) | Baseline and week 12
  Fear of movement measured with the Tampa Scale. Higher scores indicate greater kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jaén, Jaén, JAEN, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be available on reasonable request to the corresponding author after publication and for 5 years, in accordance with data protection policies.
Supporting Information: Study Protocol, ICF
Time Frame: From 6 months after publication
Access Criteria: Requests with a brief proposal; data use agreement required.
URL: https://www.ujaen.es/departamentos/ciesal/contactos/cruz-diaz-david